CLINICAL TRIAL: NCT05643508
Title: A Randomized, Double-blind, Multicenter Phase 3 Trial to Evaluate the Efficacy and Safety of Co-administration of DWC202206 and DWC202207 in Patients With Hypertension and Dyslipidemia
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of DWC202206 and DWC202207 in Patients With Concomitant Hypertension and Hyperlipidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1575301
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (D) DWC202206 + DWC202207 (Experimental)
  Interventions: Drug: (D) DWC202206; Drug: (D) DWC202207
- (P+D) DWC202206 + DWC202207 (Active Comparator)
  Interventions: Drug: (D) DWC202207; Drug: (P) DWC202206
- (D+P) DWC202206 + DWC202207 (Active Comparator)
  Interventions: Drug: (D) DWC202206; Drug: (P) DWC202207

INTERVENTIONS:
Drug: (D) DWC202206 — Drug of DWC202206 A mg
  Arms: (D) DWC202206 + DWC202207; (D+P) DWC202206 + DWC202207
Drug: (D) DWC202207 — Drug of DWC202207 B/C mg
  Arms: (D) DWC202206 + DWC202207; (P+D) DWC202206 + DWC202207
Drug: (P) DWC202206 — Placebo of DWC202206 A mg
  Arms: (P+D) DWC202206 + DWC202207
Drug: (P) DWC202207 — Placebo of DWC202207 B/C mg
  Arms: (D+P) DWC202206 + DWC202207

SUMMARY:
This study aims to evaluate the efficacy and safety of co-administration of DWC202206 and DWC202207 in patients with concomitant hypertension and hyperlipidemia.

DETAILED DESCRIPTION:
The study design is a randomized, double-blind, multicenter clinical trial. The patients were randomly assigned to each group. Primary endpoint was the change of MSSBP based on baseline between Treatment arm and control 1 arm and the change of LDL-C based on baseline between arm and control 2 arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 80 years
* Patients with hypertension and hyperlipidemias

Exclusion Criteria:

* Orthostatic hypotension
* History of ventricular tachycardia, atrial fibrillation
* Uncontrolled diabetes mellitus

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The change of MSSBP (Mean Sitting Systolic Blood Pressure) based on baseline between treatment arm and control 1 arm | 8 weeks
The change of LDL-C based on baseline between treatment arm and control 2 arm | 8 weeks

SECONDARY OUTCOMES:
The change of MSSBP (Mean Sitting Systolic Blood Pressure) based on baseline between treatment arm and control 1 arm | 4 weeks
The change of LDL-C based on baseline between treatment arm and control 2 arm | 4 weeks